CLINICAL TRIAL: NCT02990689
Title: Clinical Study to Evaluate the Visual Performance of Three Multifocal IOLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LISA tri 839MP HEN 301-11
Record Dates: First submitted 2016-12-06; First posted 2016-12-13 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 809M (Active Comparator): bifocal intraocular lens (IOL)
  Interventions: Device: Bifocal Intraocular Lens
- 839MP (Active Comparator): trifocal intraocular lens (IOL)
  Interventions: Device: Trifocal Intraocular Lens
- SN6AD1 (Active Comparator): bifocal intraocular lens (IOL)
  Interventions: Device: Low Addition Bifocal Intraocular Lens

INTERVENTIONS:
Device: Trifocal Intraocular Lens — bifocal intraocular lens (IOL)
  Arms: 839MP
Device: Bifocal Intraocular Lens — trifocal intraocular lens (IOL)
  Arms: 809M
Device: Low Addition Bifocal Intraocular Lens — low near addition intraocular lens (IOL)
  Arms: SN6AD1

SUMMARY:
The purpose of this study is to compare the performances of 2 bifocal IOLs and 1 trifocal IOL for far, near and intermediate vision.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any gender, aged 50 to 80 years
* Signed informed consent form
* Healthy eyes besides cataract
* Assured follow-up examinations
* Stable corneal conditions within the last 12 months
* Corneal astigmatism less than 1D
* Implantation into the capsular bag by injector

Exclusion Criteria:

* Degenerative visual disorders (e.g. macular degeneration, optic nerve atrophy, or retinal disorders)
* Pseudophakia
* Cornea guttata; keratoplasty
* Irregular astigmatism (e.g. Keratoconus)
* Corneal scarring
* Diabetic retinopathy
* Aniridia
* Amblyopia
* Amotio operation; anamnesis with vitreous surgery
* Pseudoexfoliation Syndrome; Uveitis
* Previous intraocular and corneal surgery
* Intraocular tumours; endotamponade
* Glaucoma or IOP higher than 24mmHg
* Phlogistic intraocular processes or other pre-existing processes that permanently limit the best corrected visual acuity to > 0.3 logMAR
* Need for a dioptre out of the range of +16.0D to +26.0D
* Inability to achieve secure lens placement in the capsular bag
* Any other pathology or condition presenting, according to the investigator opinion, a risk for the patient
* Intraoperative complications, damaged posterior bag, intraocular haemorrhage, can opener rhexis
* Pregnancy or lactation period for female patients

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Intermediate visual acuity | 12 months

SECONDARY OUTCOMES:
Distance visual acuity | 12 months
Near visual acuity | 12 months